CLINICAL TRIAL: NCT01490372
Title: Is Gestational Diabetes Mellitus (GDM) an Independent Risk Factor for Cardiometabolic Syndrome in Offspring?
Brief Title: Gestational Diabetes Mellitus and Cardiometabolic Syndrome in Offspring
Acronym: DG3
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, endocrinologist, researcher, Université de Sherbrooke
Other Study IDs: 10-207
Record Dates: First submitted 2011-11-17; First posted 2011-12-13 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GDM offspring: Children born from gestational diabetes mellitus pregnancy
- No-GDM offspring: Children born from a normal pregnancy

SUMMARY:
Gestational Diabetes Mellitus (GDM) has long been known as leading to macrosomias, neonatal hypoglycemias and other complications which are treatable and preventable. Nowadays, GDM is recognized as an entity with long-term serious sequels to the mother (GDM is considered a forerunner of type 2 diabetes) and her offspring. Indeed, according to the programming hypothesis, GDM sets the stage for metabolic syndrome, obesity, type 2 diabetes and hypertension. However, these cross-sectional studies failed to control for maternal disease history and genetic background although heredity is a major epidemiology risk factor of type 2 diabetes. Also, studies usually refer to traditional markers such as BMI, blood pressure, lipids profile and oral glucose tolerance test (OGTT); none explored inflammatory biomarkers and adipokines in-depth, despite the possible link between their presence and the development of metabolic and cardiovascular diseases in GDM offsprings.

Exclusion of genetic confounding factors will help establish the role of GDM as an independent marker of cardiometabolic risk in GDM offspring. It is highly relevant to identify GDM as a risk factor for cardiometabolic diseases, given the worldwide obesity epidemic, the alarming prevalence increase of GDM and its serious sequels to both mother and offspring.

ELIGIBILITY:
Inclusion Criteria:

* age 4 to 12 years
* Tanner stage < 2
* to understand French or English

Exclusion Criteria:

* Type 1 diabetes
* weight < 10 kg
* placenta abnormalities
* gestational age < 34 weeks
* illness affecting growth and metabolism
* taking medications

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Offspring born from GDM pregnancies and their siblings born to the same mothers but from non-GDM pregnancies.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome | 4 to 12 years after birth.
  Prevalence of metabolic syndrome

SECONDARY OUTCOMES:
Inflammatory markers | Assessed only once 4 to 12 years after birth
  4 to 12 years after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ardilouze, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche clinique Étienne-Le Bel du CHUS, Sherbrooke, Quebec, Canada